CLINICAL TRIAL: NCT01423864
Title: Retrospective Study of Intrapleural Methylprednisolone Injection for Multiple Organ Failure With Acute Respiratory Distress Syndrome
Brief Title: Intrapleural Methylprednisolone Injection for Multiple Organ Failure With Acute Respiratory Distress Syndrome
Acronym: IP steroid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200906014R
Record Dates: First submitted 2011-08-18; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Multiple Organ Failure
Keywords: Acute Respiratory Distress Syndrome; Multi-organ Dysfunction Syndrome; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome; Multiple Organ Failure | interventions — hydrocortisone hemisuccinate; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional ECMO with intravenous steroid (Sham Comparator): refractory acute respiratory distress syndrome and multi-organ dysfunction syndrome unresponsive to conventional extracorporeal membrane oxygenation
  Interventions: Drug: conventional ECMO with intravenous steroid
- Drug: intrapleural steroid instillation (Experimental): refractory acute respiratory distress syndrome and multi-organ dysfunction syndrome unresponsive to conventional extracorporeal membrane oxygenation
  Interventions: Drug: solumedrol

INTERVENTIONS:
Drug: conventional ECMO with intravenous steroid — refractory acute respiratory distress syndrome and multi-organ dysfunction syndrome treated with intravenous steroid, Solu-Cortef 50mg q6h taper down when hemodynamic stable
  Other Names: Solu-Cortef
  Arms: conventional ECMO with intravenous steroid
Drug: solumedrol — Initially, intrapleural steroid administration was performed using 40 mg solumedrol q6h (for both the pleural cavities). If chest radiography showed an improvement in consolidation, i.e., 0.8 > FiO2 ≥ 0.5 and 5 ≤ PEEP ≤ 10, the dosage of solumedrol was reduced to 40 mg q12h. When FiO2 was below 0.5 and the PEEP was below 10, the dosage of solumedrol was lowered to 40 mg qd for 3 days and then its administration was discontinued.
  Arms: Drug: intrapleural steroid instillation

SUMMARY:
Acute respiratory distress syndrome (ARDS) in combination with multi-organ dysfunction syndrome (MODS) is a life-threatening condition, particularly when treatment modalities such as extracorporeal membrane oxygenation (ECMO) and catecholamine administration have failed to treat the severe condition. In this study, the investigators report patients who responded to intrapleural steroid instillation (IPSI) while being unresponsive to conventional treatment (use of intravenous steroids, nitric oxide inhalation, high-frequency oscillatory ventilation, or ECMO) for treatment of critical illnesses such as ARDS in combination with MODS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) with multi-organ dysfunction syndrome (MODS) are common debilitating postoperative complications, which also result from shock and trauma. However, despite the use of ECMO, mortality rate among hypoxia patients remains high in such critical care conditions. Corticosteroid therapy inhibits ongoing inflammation and abnormal deposition of collagen. However, intravenous administration of corticosteroids may be harmful because it may increase the risk of associated neuromyopathy in critically ill patients. Although intrapleural instillation of steroids has been employed in several pleural diseases,little is known about the therapeutic effects of this treatment method on ARDS in combination with MODS. Therefore, in the present pilot study, the investigators hypothesized that timely initiation of intrapleural steroid instillation (IPSI) will positively influence ventilation in and survival of patients with ARDS in combination with MODS.

The investigators conducted a retrospective study on ninety-two of the 467 ECMOs performed between 2005 and 2009 were on ARDS patients. Analyses of gas exchange, tidal volumes, airway pressures, respiratory frequency, and vasopressor and sedation requirements were performed before and after intervention.

The indication for IPSI was unresponsive severe ARDS in combination with MODS when all the other treatment modalities such as intravenous steroid administration, nitric oxide inhalation, high-frequency oscillatory ventilation, or ECMO performed within 2 days were unsuccessful.

An experienced team performed thoracic catheterization of the patients under ultrasound evaluation. Patients with severe pleural adhesion were considered unsuitable for IPSI. The dosage of the intrapleural steroid was determined on the basis of the chest radiographic examination, inspired oxygen concentration, and positive end-expiratory pressure (PEEP) of the ventilator.

ELIGIBILITY:
Inclusion Criteria:

1. All of the patients had failure of at least 2 organs acquiring arteriovenous or venovenous ECMO support
2. All of the patients met the criteria as below:

   * blood gas parameters of PaO2/FiO2 < 100
   * bilateral pulmonary infiltration on chest radiographic images
   * 100% oxygen demand in case of ventilation and ECMO flow
   * hemodynamic instability requiring high catecholamine infusion
   * All the patients had scoring system, which were calculated by the physician within 24 h of admission of the patients into the hospital.

     * sequential organ failure assessment score (SOFA) ≥ 10
     * Acute Physiology and Chronic Health Evaluation II (APACHE II) score ≥ 20
     * inotropic score ≥ 10
     * multiple organ dysfunction (MOD) score ≥ 10

Exclusion Criteria:

1. uncontrollable underlying disease
2. life expectancy of less than 24 h
3. immunosuppression
4. neutrophil count of less than 0.3 × 109/L
5. brainstem death
6. history of long-term corticosteroid use during the past 6 months.

Ages: 16 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
survival until discharge from the hospital | 2005~2009 (up to 4 years)
  Comparing the difference between two groups about the survival ratio of discharge from the hospital

SECONDARY OUTCOMES:
Incidence of complications | 12 weeks
  complication of the interventional treatment will be followed for the duration of hospital stay
the effects on tidal volumes | up to 12 weeks
  the therapeutic effects in the improvement of tidal volumes, followed for the duration of ventilator usage
the therapeutic effects on oxygenation | up to 12 weeks
  the therapeutic effects in the improvement of oxygenation, followed for the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ming Huang, MD, MS, Principal Investigator — National Taiwan University Hospital and National Taiwan University College of Medicine
Locations (1):
- Department of Surgery, National Taiwan University Hospital, 7, Chung-Shan S. Rd, Taipei 10002, Taiwan., Taiwan, Taiwan

REFERENCES:
- [Background] Zhang J, Wang W, Sun J, Li Q, Liu J, Zhu H, Chen T, Wang H, Yu S, Sun G, Chen W, Yi D. Gap junction channel modulates pulmonary vascular permeability through calcium in acute lung injury: an experimental study. Respiration. 2010;80(3):236-45. doi: 10.1159/000274384. Epub 2010 Jan 7. PMID 20090287
- [Background] Suchyta MR, Clemmer TP, Orme JF Jr, Morris AH, Elliott CG. Increased survival of ARDS patients with severe hypoxemia (ECMO criteria). Chest. 1991 Apr;99(4):951-5. doi: 10.1378/chest.99.4.951. PMID 2009801
- [Background] Biffl WL, Moore FA, Moore EE, Haenel JB, McIntyre RC Jr, Burch JM. Are corticosteroids salvage therapy for refractory acute respiratory distress syndrome? Am J Surg. 1995 Dec;170(6):591-5; discussion 595-6. doi: 10.1016/s0002-9610(99)80022-1. PMID 7492007
- [Background] Brunet F, Mira JP, Belghith M, Monchi M, Renaud B, Fierobe L, Hamy I, Dhainaut JF, Dall'ava-Santucci J. Extracorporeal carbon dioxide removal technique improves oxygenation without causing overinflation. Am J Respir Crit Care Med. 1994 Jun;149(6):1557-62. doi: 10.1164/ajrccm.149.6.8004313.
- [Background] Wiener-Kronish JP, Broaddus VC. Interrelationship of pleural and pulmonary interstitial liquid. Annu Rev Physiol. 1993;55:209-26. doi: 10.1146/annurev.ph.55.030193.001233. PMID 8466174
- [Background] Lewandowski K, Rossaint R, Pappert D, Gerlach H, Slama KJ, Weidemann H, Frey DJ, Hoffmann O, Keske U, Falke KJ. High survival rate in 122 ARDS patients managed according to a clinical algorithm including extracorporeal membrane oxygenation. Intensive Care Med. 1997 Aug;23(8):819-35. doi: 10.1007/s001340050418. PMID 9310799
- [Background] Dagenais A, Denis C, Vives MF, Girouard S, Masse C, Nguyen T, Yamagata T, Grygorczyk C, Kothary R, Berthiaume Y. Modulation of alpha-ENaC and alpha1-Na+-K+-ATPase by cAMP and dexamethasone in alveolar epithelial cells. Am J Physiol Lung Cell Mol Physiol. 2001 Jul;281(1):L217-30. doi: 10.1152/ajplung.2001.281.1.L217. PMID 11404265
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] North SA, Au HJ, Halls SB, Tkachuk L, Mackey JR. A randomized, phase III, double-blind, placebo-controlled trial of intrapleural instillation of methylprednisolone acetate in the management of malignant pleural effusion. Chest. 2003 Mar;123(3):822-7. doi: 10.1378/chest.123.3.822. PMID 12628884
- [Background] Gerlach H, Keh D, Semmerow A, Busch T, Lewandowski K, Pappert DM, Rossaint R, Falke KJ. Dose-response characteristics during long-term inhalation of nitric oxide in patients with severe acute respiratory distress syndrome: a prospective, randomized, controlled study. Am J Respir Crit Care Med. 2003 Apr 1;167(7):1008-15. doi: 10.1164/rccm.2108121. PMID 12663340
- [Background] Broccard AF. Prone position in ARDS: are we looking at a half-empty or half-full glass? Chest. 2003 May;123(5):1334-6. doi: 10.1378/chest.123.5.1334. No abstract available. PMID 12740242
- [Background] Dunser M, Hasibeder W, Rieger M, Mayr AJ. Successful therapy of severe pneumonia-associated ARDS after pneumonectomy with ECMO and steroids. Ann Thorac Surg. 2004 Jul;78(1):335-7. doi: 10.1016/S0003-4975(03)01264-5. PMID 15223462
- [Background] Tomiyama H, Takara I, Tokumine J, Sugahara K. [Sivelestat sodium hydrate was effective for ARDS in a patient suffering from chronic rheumatoid arthritis with acute exacerbation after failing to respond to high dose steroid pulse therapy]. Masui. 2004 Sep;53(9):1042-6. Japanese. PMID 15500109
- [Background] Zemans RL, Matthay MA. Bench-to-bedside review: the role of the alveolar epithelium in the resolution of pulmonary edema in acute lung injury. Crit Care. 2004 Dec;8(6):469-77. doi: 10.1186/cc2906. Epub 2004 Jun 30. PMID 15566618
- [Background] Shinozaki M. [Respiratory and cadiovascular management of septic ALI-ARDS and shock]. Nihon Rinsho. 2004 Dec;62(12):2301-7. Japanese. PMID 15597800
- [Background] Lee HS, Lee JM, Kim MS, Kim HY, Hwangbo B, Zo JI. Low-dose steroid therapy at an early phase of postoperative acute respiratory distress syndrome. Ann Thorac Surg. 2005 Feb;79(2):405-10. doi: 10.1016/j.athoracsur.2004.07.079. PMID 15680804
- [Background] Bernard GR. Acute respiratory distress syndrome: a historical perspective. Am J Respir Crit Care Med. 2005 Oct 1;172(7):798-806. doi: 10.1164/rccm.200504-663OE. Epub 2005 Jul 14. PMID 16020801
- [Background] Annane D, Sebille V, Bellissant E; Ger-Inf-05 Study Group. Effect of low doses of corticosteroids in septic shock patients with or without early acute respiratory distress syndrome. Crit Care Med. 2006 Jan;34(1):22-30. doi: 10.1097/01.ccm.0000194723.78632.62. PMID 16374152
- [Background] Beiderlinden M, Eikermann M, Boes T, Breitfeld C, Peters J. Treatment of severe acute respiratory distress syndrome: role of extracorporeal gas exchange. Intensive Care Med. 2006 Oct;32(10):1627-31. doi: 10.1007/s00134-006-0262-y. Epub 2006 Jul 28. PMID 16874497